CLINICAL TRIAL: NCT00073359
Title: Engagement and Alliance in CBT for Depressed Adolescents
Brief Title: Effects of Therapist Behavior on the Treatment of Depressed Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21MH065988 (NIH); R21MH065988 (NIH); DSIR CT-S
Record Dates: First submitted 2003-11-19; First posted 2003-11-21 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Depression; Depressive Disorder; Dysthymic Disorder
Keywords: Adolescent
MeSH Terms: conditions — Depression; Depressive Disorder; Dysthymic Disorder | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy

SUMMARY:
The purpose of this study is to identify and evaluate therapist behaviors that affect how well and how long adolescent patients stay in treatment for depression.

DETAILED DESCRIPTION:
Early patient drop out, sporadic attendance, and minimal participation have hindered the development and administration of effective treatments for adolescent depression. Adolescents who do not receive adequate exposure to active treatment are unlikely to benefit from experimentally supported treatments. Certain therapist behaviors may influence the attendance, drop-out, and overall participation of adolescents with depression. This study will evaluate the effect of engagement interventions and alliance on attendance, participation, completion, and outcome in depressed adolescents.

Participants in this study will have 12 weekly sessions of cognitive behavioral therapy (CBT) at a school-based health clinic. Audio recordings from the completed CBT sessions will be replayed and evaluated to identify therapist engagement interventions, therapy alliance, and treatment participation.

ELIGIBILITY:
Inclusion Criteria:

* Major depression or dysthymic disorder
* Referred by school

Exclusion Criteria:

* Comorbid psychosis, bipolar disorder, or mental retardation

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2003-02; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Denver Public Schools Health Clinics, Denver, Colorado, United States